CLINICAL TRIAL: NCT02557607
Title: Quantification of Cerebral Blood Flow by Arterial Spin Labeling in the Screening and Monitoring of Vasospasm in Subarachnoid Haemorrhage
Brief Title: Quantification of Cerebral Blood Flow by Arterial Spin Labeling in Vasospasm in Subarachnoid Haemorrhage
Acronym: ASL-HSA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CHU-P 2013-06
Record Dates: First submitted 2015-09-18; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monitoring a subarachnoid hemorrhage (Other): Any patient hospitalized at the University Hospital of Angers in neurosurgical intensive care unit for supervision by ASL and DTC a subarachnoid hemorrhage from all etiologies (excluding traumatic). An analysis of the three sessions MRI performed systematically within the first 14 days of the start of symptoms revealing the HSA will be
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — An analysis of the three sessions MRI performed systematically within the first 14 days of the start of symptoms revealing the HSA will be

SUMMARY:
A technique of MRI infusion -l'Arterial Spin Labeling-, non-invasive and non-irradiating, repeatable over time, appears promising in the field. This sequence allows for routine, generate perfusion maps relating to the entire brain volume

DETAILED DESCRIPTION:
The subarachnoid hemorrhage (SAH) is a relatively severe disease whose prognosis is particularly related to the early onset of arterial vasospasm, maximum between the 5th and 14th day after SAH. Many obstacles make it difficult screening and monitoring of such complication. The challenge is to be able to demonstrate a reduction in regional cerebral blood flow before the onset of irreversible parenchymal sequelae, responsible for the majority of long-term morbidity among survivors. In clinical routine, screening vasospasm is achieved by Doppler intracranial arteries (DTC). However, its sensitivity is poor with regard to the middle and anterior cerebral arteries. The gold standard for diagnosis is cerebral arteriography. However, vasospasm in arteriography or trans-cranial Doppler does not prejudice the appearance of a delayed ischemic deficit.

A technique of MRI infusion -l'Arterial Spin Labeling-, non-invasive and non-irradiating, repeatable over time, appears promising in the field. This sequence allows for routine, generate perfusion maps relating to the entire brain volume

ELIGIBILITY:
Inclusion Criteria:

* Adults.
* Who have given their written consent.
* Affiliated to a social security system.
* Any patient hospitalized at the University Hospital of Angers in neurosurgical intensive care unit for supervision by ASL and DTC a subarachnoid hemorrhage from all etiologies (excluding traumatic).

Exclusion Criteria:

* Contraindications to MRI
* patient hospitalized at the University Hospital of Angers in surgical intensive care for monitoring a subarachnoid hemorrhage.
* patient hospitalized at the University Hospital of Angers for monitoring a subarachnoid hemorrhage traumatic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
exploitation of raw images provided with the waning of the acquisition of the sequence ASL. | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Aram TER MINASSIAN, Physician, Principal Investigator — UH ANGERS
Locations (1):
- CHU Angers, Angers, France